CLINICAL TRIAL: NCT02496650
Title: Dexmedetomidine Addition to Benzodiazepines for Patients With Alcohol Withdrawal Syndrome in the ICU: a Randomised Controlled Study
Brief Title: Dexmedetomidine Addition to Benzodiazepines for Patients With Alcohol Withdrawal State in the ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Kateryna Bielka, Medical doctor, clinical resident, Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 234
Record Dates: First submitted 2015-07-10; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Alcohol Withdrawal State
Keywords: alcohol withdrawal state; dexmedetomidine; benzodiasepines; intensive care
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group D (Experimental): Dexmedetomidine (DEX) infusion was started in doses 0,2-1,4 μg/kg/hr and titrated to achieve target sedation level; symptom-triggered BZD administration (diazepam 10mg bolus) were used wherever DEX infusion was not enough. Antipsychotics (haloperidol 5mg boluses) were used as a rescue medication for severe agitation or hallucinations.
  Interventions: Drug: Dexmedetomidine
- Group C (No Intervention): Benzodiasepine (BZD) boluses (diazepam 10mg) were used to achieve target sedation level and to control AWS symptoms (symptom-triggered administration). Antipsychotics (haloperidol 5mg boluses) were used as a rescue medication for severe agitation or hallucinations.

INTERVENTIONS:
Drug: Dexmedetomidine — DEX infusion in doses 0,2-1,4 μg/kg/hr
  Other Names: Dexdor
  Arms: Group D

SUMMARY:
The objective of this randomized controlled study was to evaluate whether DEX addition to benzodiazepine therapy is effective and safe for AWS patients in the intensive care unit (ICU). Eligible participants were randomly assigned to intervention (D) and control (C) groups. In the group D DEX infusion was started in doses 0,2-1,4 μg/kg/hr and titrated to achieve target sedation level; symptom-triggered BZD administration (diazepam 10mg bolus) were used wherever DEX infusion was not enough. In group K BZD boluses (diazepam 10mg) were used to achieve target sedation level and to control AWS symptoms (symptom-triggered administration). The primary efficacy outcomes were 24-hour diazepam consumption and cumulative diazepam dose required over the course of ICU stay, secondary outcomes were length of ICU stay, sedation and communication quality, haloperidol consumption.

DETAILED DESCRIPTION:
Ethical issues This study was approved by the Bogomolets National Medical University ethics committee and a written informed concern was obtained from the patient, the patient's family or a legal representative.

Study design This randomized, single-center, controlled study was conducted in the adult ICU at private hospital "Boris" in Kiyv (Ukraine). The inclusion criteria were: age 18 or older, signed informed concern, within 2 hours of ICU admission, diagnosed alcohol withdrawal syndrome or alcohol withdrawal delirium by DSM IV criteria (). The exclusion criteria were age younger than 18 or older than 75, history of use or withdrawal states of other psychoactive substances, general anesthesia during last 24 hours or known other sedatives use, severe neurologic disorder (traumatic brain injury, acute stroke, severe dementia), pregnancy or lactation, severe comorbidities (severe heart failure, acute myocardial infarction, heart rate <50/min, glomerular filtration rate < 30 ml/min, liver failure Child-Pugh class C), known allergy to the study medication.

After primary patient assessment the target sedation level was set individually and study treatment begun. Eligible participants were randomly assigned in a 1:1 ratio to the intervention (group D) and control groups using random assignment in block of four. In group D DEX infusion was started in doses 0,2-1,4 μg/kg/hr and titrated to achieve target sedation level; symptom-triggered BZD administration (diazepam 10mg bolus) were used wherever DEX infusion was not enough. In group K BZD boluses (diazepam 10mg) were used to achieve target sedation level and to control AWS symptoms (symptom-triggered administration). Antipsychotics (haloperidol 5mg boluses) were used as a rescue medication in both groups for severe agitation or hallucinations.

Study outcomes and statistical analysis The primary efficacy outcomes were 24-hour diazepam consumption after study begins and cumulative diazepam dose required over the course of ICU stay.

The secondary efficacy outcomes include:

* length of ICU stay and intubation rates;
* sedation quality: the time of target sedation (proportion of time in target sedation range (in most cases RASS score 0 to -2) to the total sedation time); the time of insufficient sedation (duration of ineffective sedation (in most cases RASS score ≥+2) to the total sedation time); the time of oversedation (duration of excessive sedation (in most cases RASS ≤-3) to the total sedation time); the number of rescue sedation boluses and sedation stops in 24 hours;
* communication quality (from 0 to 10, were 0 - uncommunicative, 10 - patient communicates well) and ability to asses pain with Visual Analogue Scale (VAS);
* haloperidol requirements and cumulative dose during ICU stay. Safety was estimate by monitoring vital sighs, ECG, laboratory tests (paO2, SaO2, blood sugar), and adverse events. Adverse events were evaluated if systolic blood pressure was lower than 90 mm Hg of higher than 160 mm Hg or heart rate was lower than 50/min or higher than 110/min; desaturation were estimated as SpO2 (or SaO2) lower than 90%; hypoglycemia was defined as serum glucose lower than 4 mmol/L and hyperglycemia as higher than 10 mmol/L. Intervention for bradycardia, tachycardia, hypertension and hypotension were titration or interruption of study agent or drug therapy.

Sedation was assessed using Richmond Agitation Sedation Scale (RASS) and AWS symptoms severity - with Clinical Institute Withdrawal Assessment of Alcohol Scale, Revised (CIWA-Ar). RASS was monitored every 2-6 hours and prior to rescue therapy, CIWA-Ar was assessed on the daily basis during sedation stops.

Randomization sequence was generated using a computer algorithm [www.random.org]. Both randomization and data analysis were conducted by independent blind member of research team.

A statistical analysis was performed using Statistics 6.0 and R software. Categorical data are presented as proportions; continuous data - as medians (InterQuartile Range, IQR 25-75%). Chi-square testing demonstrates that all variables under study are discrete. To assess significances two-tailed Mann-Whitney U test and Fisher exact test were used. A P-value of less than 0.05 defined as significant.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older,
* signed informed concern,
* within 2 hours of ICU admission,
* diagnosed alcohol withdrawal syndrome or alcohol withdrawal delirium by DSM IV criteria

Exclusion Criteria:

* younger than 18 or older than 75,
* history of use or withdrawal states of other psychoactive substances,
* general anesthesia during last 24 hours or known other sedatives use,
* severe neurologic disorder (traumatic brain injury, acute stroke, severe dementia),
* pregnancy or lactation,
* severe comorbidities (severe heart failure, acute myocardial infarction, heart rate <50/min, glomerular filtration rate < 30 ml/min, liver failure Child-Pugh class C),
* known allergy to the study medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
24-hour diazepam consumption | 24 hours
  24-hour diazepam consumption was estimated after the study begins.
Cumulative diazepam dose | 30 days
  Diazepam dose required over the course of ICU stay

SECONDARY OUTCOMES:
Length of ICU stay | 30 days
the time of target sedation | 24 hours
  proportion of time in target sedation range (in most cases RASS score 0 to -2) to the total sedation time
the number of rescue sedation boluses | 24 hours
the number of sedation stops | 24 hours
Adverse events | 30 days
  hypotension, hypertension, tachycardia, bradicardia, desaturation

REFERENCES:
- [Derived] Bielka K, Kuchyn I, Glumcher F. Addition of dexmedetomidine to benzodiazepines for patients with alcohol withdrawal syndrome in the intensive care unit: a randomized controlled study. Ann Intensive Care. 2015 Dec;5(1):33. doi: 10.1186/s13613-015-0075-7. Epub 2015 Nov 2. PMID 26525052